CLINICAL TRIAL: NCT03560479
Title: A Randomized Placebo Controlled Phase I/II Study Evaluating the Safety and Efficacy of alpha1H in Adult Patients With Non-muscle Invasive Bladder Cancer Awaiting Transurethral Surgery
Brief Title: A First-in-Human Study of alpha1H in Patients With Non-muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamlet Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP002-001; 2016-004269-14 (EudraCT Number)
Record Dates: First submitted 2018-05-24; First posted 2018-06-18 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: First-in human; Phase 1; Phase 2; Safety; Tolerability; Cancer; Bladder cancer; Clinical trial; Anti-cancer; Antineoplastic; alpha1H; HAMLET; Urothelial; Malignant; Papillary; Transurethral; Non-muscle invasive; Instillation; Intravesical
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Part 1 (Main part): Patients are randomized to receive intravesical instillations of either alpha1H (7.4 mg/mL) or placebo. The randomization ratio is 1:1.
  Part 2 (DE part): In this open part of the study, two groups of patients will receive escalating doses of alpha1H in a standard 3+3 design. One group will receive a dose of 37 mg/mL and, if tolerated, one group will receive a dose of 74 mg/mL.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- alpha1H, 7.4 mg/mL (Experimental): alpha1H (7.4 mg/mL), solution for instillation, 30 mL
  Interventions: Drug: alpha1H, 7.4 mg/mL
- placebo (Placebo Comparator): Placebo, 0.9% NaCl (sodium chloride), 30 mL
  Interventions: Other: placebo
- alpha1H, 37 mg/mL (Experimental): alpha1H (37 mg/mL), solution for instillation, 30 mL
  Interventions: Drug: alpha1H, 37 mg/mL
- alpha1H, 74 mg/mL (Experimental): alpha1H (74 mg/mL), solution for instillation, 30 mL
  Interventions: Drug: alpha1H, 74 mg/mL

INTERVENTIONS:
Drug: alpha1H, 7.4 mg/mL — Intravesical instillations on 6 occasions during 22 days (Days 1, 3, 5, 8, 15 and 22)
  Arms: alpha1H, 7.4 mg/mL
Other: placebo — Intravesical instillations on 6 occasions during 22 days (Days 1, 3, 5, 8, 15 and 22)
  Arms: placebo
Drug: alpha1H, 37 mg/mL — Intravesical instillations on 6 occasions during 22 days (Days 1, 3, 5, 8, 15 and 22)
  Arms: alpha1H, 37 mg/mL
Drug: alpha1H, 74 mg/mL — Intravesical instillations on 6 occasions during 22 days (Days 1, 3, 5, 8, 15 and 22)
  Arms: alpha1H, 74 mg/mL

SUMMARY:
This study evaluates the tolerability and preliminary anti-tumour effect of alpha1H in adults with non-muscle invasive bladder cancer, who are awaiting transurethral surgery.

In the main, blinded part of the study, one group of subjects will receive treatment with alpha1H and the other half will receive placebo. In a second, dose-escalation part of the study, a third and fourth group of subjects will receive increased doses of alpha1H.

The treatment is given on 6 occasions during a period of 22 days. The study duration is 8 - 12 weeks including scheduled follow-up and up to 27 months when an optional 24-months non-interventional follow-up period is included.

DETAILED DESCRIPTION:
Protein-lipid complexes represent a new type of tumouricidal biologicals, with broad effects against cancers of different origins. The investigational product alpha1H is a synthetic peptide, corresponding to the alpha1 domain of α-lactalbumin, in complex with oleic acid. Alpha1H is a further development product of HAMLET, a complex between human alpha-lactalbumin and oleic acid, which has shown broad anti-tumor activity with a high degree of selectivity.

This study is a combined phase 1/2, placebo controlled, double blind study in subjects with non-muscle invasive bladder cancer awaiting transurethral resection of bladder (TURB). The first, main part of the study is randomized 1/1 and the subjects will receive intravesical instillation of either alpha1H or placebo on 6 occasions during a period of 22 days (on days 1, 3, 5, 8, 15 and 22). In a second, open, dose-escalation (DE) part of the study, two additional groups will receive increased doses of alpha1H in a standard 3+3 design in order to determine a Maximum Tolerated Dose (MTD) or alternatively, a Maximum Administered Dose (MAD). The same treatment schedule as in part 1 will be followed. One group will receive a dose of 5 times the original dose and, if tolerated, the last group will receive a dose of 10 times the original dose.

Cell shedding is quantified and characterized at each treatment occasion. The bladder tumors are characterized prior treatment and prior to the scheduled surgery. Remaining tumors will be removed by TURB (according to European Association of Urology (EAU) Guidelines recommendations) and tissues will be obtained for analyses.

A follow-up Visit will take place 30 days after the last administration of study treatment.

The total study duration of the main study is 8 - 12 weeks. After the main study, the subjects may continue in an optional extended 24-months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-muscle invasive papillary bladder cancer (NMIBC) based on cystoscopy appearance, on the waiting list for TURB.
* Negative pregnancy test in women of childbearing potential.
* Appropriate methods of contraception in women of childbearing potential during study.
* Patients should be able to keep the content of the bladder for at least one hour.

Exclusion Criteria:

* Patient with a previous history of muscle invasive bladder cancer.
* Patient with a history of NMIBC with an interval shorter than 6 months after previous TURB.
* Previous intravesical Bacillus Calmette-Guerin (BCG) immunotherapy in the last 12 months.
* Previous intravesical chemotherapy in the last 12 months.
* Participants with any other cancer diagnosis within the last 5 years (except of skin basaliomas).
* Acute urinary tract infection
* Participants with prior radiotherapy or systemic chemotherapy.
* Participants receiving any other investigational agent or non-marketed product one month prior to Visit 1 and during the trial.
* Any concurrent illness that may render a participant ineligible or limit compliance with study requirements.
* Previously enrolled in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety as Adverse Events Profile | From signing of informed consent (Day 1) and until 30 days after the last dose (Day 52).
  Incidence of adverse events and classification in terms of severity, causality and outcome
Efficacy as Cell Shedding | Days 1 to 22
  Change in cell shedding into urine (number of epithelial cells per mL of urine).
Change from baseline in characteristics of papillary tumors | Prior to treatment (Baseline) and on Day 30, in connection with scheduled surgery.
  The bladder tumors will be characterised by in vivo imaging during examination by cystoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Marek Babjuk, MD, Prof., Principal Investigator — Motol University Hospital
Locations (1):
- Motol University Hospital, Prague, Czechia

REFERENCES:
- [Derived] Brisuda A, Ho JCS, Kandiyal PS, Ng JT, Ambite I, Butler DSC, Hacek J, Wan MLY, Tran TH, Nadeem A, Tran TH, Hastings A, Storm P, Fortunati DL, Esmaeili P, Novotna H, Hornak J, Mu YG, Mok KH, Babjuk M, Svanborg C. Bladder cancer therapy using a conformationally fluid tumoricidal peptide complex. Nat Commun. 2021 Jun 8;12(1):3427. doi: 10.1038/s41467-021-23748-y. PMID 34103518